CLINICAL TRIAL: NCT05788393
Title: Opioid Sparing Analgesia Continuous Intraoperative Infusion of Dexmedetomidine Versus Lidocaine for Laparoscopic Cholecystectomy a Randomized Double-blind Clinical Trial
Brief Title: Opioid Sparing Analgesia Continuous Intraoperative Infusion of Dexmedetomidine Versus Lidocaine for Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Daniel Hanna, Primary investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Analgesia in cholecystectomy
Record Dates: First submitted 2023-01-17; First posted 2023-03-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2023-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: this study is to compare the effects of continuous intraoperative infusion of dexmedetomidine versus lidocaine as opioid sparing analgesia on patients undergoing laparoscopic cholecystectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): This group will receive continuous intraoperative dexmedetomidine IV infusion [1ug/kg dexmedetomidine over 15 min as a loading dose and 0.5ug/kg/h for maintenance].
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Lidocaine group (Experimental): This group will receive continuous intraoperative lidocaine IV infusion [1.5 mg/kg lidocaine over 15 min as a loading dose and 1.5 mg/kg/h for maintenance].
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — dexmedetomidine group will receive continuous intraoperative dexmedetomidine IV infusion [1ug/kg dexmedetomidine over 15 min as a loading dose and 0.5ug/kg/h for maintenance].The continuous intraoperative IV infusion of study drug will be stopped 10 min before the end the surgical procedure.
  Arms: Dexmedetomidine group
Drug: Lidocaine IV — lidocaine group will receive continuous intraoperative lidocaine IV infusion [1.5 mg/kg lidocaine over 15 min as a loading dose and 1.5 mg/kg/h for maintenance]. The continuous intraoperative IV infusion of study drug will be stopped 10 min before the end the surgical procedure.
  Arms: Lidocaine group

SUMMARY:
Opioid sparing analgesia: Continuous intraoperative infusion of dexmedetomidine versus lidocaine for laparoscopic cholecystectomy, a randomized double-blind clinical trial.

DETAILED DESCRIPTION:
Postoperative pain represents one of the most common complaints following surgeries. Despite advances in modern medicine, pain following surgical procedures is still a challenge for anesthetists, though significant progress made over the past decades. The mechanism of pain following laparoscopic procedures is thought to be multifactorial. The main causes of pain after laparoscopic cholecystectomy (LC) are pain from the incision site, pneumoperitoneum and cholecystectomy. Clinicians using different methods for analgesia after LC. like non-steroidal anti-inflammatory drugs, intraperitoneal local anesthetics, local anesthetics applied to the wound site, removal of the insufflation gas, paravertebral block (PVB), and epidural block. To date, the mainstay of management has been the administration of exogenous opioids such as morphine or fentanyl. However, pain is not always fully relieved by such agents, and often patients develop tolerance to them. The ever-increasing doses of opioids are clearly not without their adverse effects. In addition to that, many patients and even some clinicians wrongly believe that addiction can be inevitable after administration of opioids. Dexmedetomidine is an alpha 2-adrenergic agonist which is a relatively new drug used for procedural sedation. It has sedative and anxiolytic effects and is known for its analgesic potential owing to a reduction of sympathetic tone. Dexmedetomidine has dose-dependent effects, ranging from minimal to deep sedation. Moreover, except at doses that cause very deep sedation or general anesthesia, the sedation is reversible. These are unique properties among the sedative medications in common use. Dexmedetomidine does not impair the respiratory drive per se and seldom causes apnea. However, it has been shown to impair the respiratory responses to hypoxia and hypercapnia and can cause hemodynamic effects such as hypertension, hypotension and bradycardia. Systemic lidocaine has centrally and peripherally analgesic, anti-hyperalgesic and anti-inflammatory effects with reduced side-effects especially if used with appropriate dose. Recently, intravenous lidocaine infusion is considered a part of analgesic therapy regimen that decreases postoperative opioid requirements and enhances convalescence after major surgeries. Dexmedetomidine and lidocaine are common adjuvant medicine anesthetics during operation for the sedative and analgesic properties. Besides, some studies have proved that both are effective in relieving postoperative pain in adults. However, there are very limited studies comparing the effects of the two adjuvant analgesics on postoperative pain in patients undergoing laparoscopic cholecystectomy (LC).

ELIGIBILITY:
Inclusion Criteria:

* Patient's status ASA status-I and II.
* Patients age above 18 years old.
* Patients scheduled for laparoscopic cholecystectomy.

Exclusion Criteria:

* Patient refusal.
* Patients with known allergy to dexmedetomidine or lidocaine.
* Patients with significant hepatic dysfunction.
* Patients with severe renal disease.
* Patients with chronic pain.
* Regular use analgesics, antidepressants or opioids in last month.
* Any known convulsive disorder.
* Significant heart disease.
* Morbid obesity (BMI>35).
* Patients with autoimmune disease
* Patients on corticosteroid therapy
* Pregnancy
* Breast feeding
* Woman under hormonal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 15 minutes
  Numeric Pain Rating Scale (NPRS) will be explained to the patient to be able to choose the score that best expressed the intensity of pain postoperatively ranging from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable".

SECONDARY OUTCOMES:
Richmond Agitation-Sedation Scale | 15 minutes
  Richmond Agitation-Sedation Scale (RASS) will be used to evaluate the level of sedation in post-anesthesia care unit (PACU), It is a 10-point scale, with four levels of anxiety or agitation, one level denoting a calm and alert state, and 5 levels of sedation, ranging from +4 to -5, desirable score is 0 to -2.
First call for rescue analgesic (Nalbuphine) | 1 day
The total postoperative Nalbuphine consumption | 1 day
Intraoperative automated non-invasive blood pressure monitoring. | 1 hour
Intraoperative electrocardiogram (ECG) heart rate monitoring. | 1 hour
The mean duration of PACU stay. | 3 hours

OTHER OUTCOMES:
Side effects of study drugs. | 1 hour
Satisfaction of the patients questionnaire | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S. Saad, Dr, Principal Investigator — Assiut university hospitals
Locations (1):
- Assiut university hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitra S, Carlyle D, Kodumudi G, Kodumudi V, Vadivelu N. New Advances in Acute Postoperative Pain Management. Curr Pain Headache Rep. 2018 Apr 4;22(5):35. doi: 10.1007/s11916-018-0690-8. PMID 29619627
- [Background] Meera A. Pain and Opioid Dependence: Is it a Matter of Concern. Indian J Palliat Care. 2011 Jan;17(Suppl):S36-8. doi: 10.4103/0973-1075.76240. PMID 21811368
- [Background] Barends CR, Absalom A, van Minnen B, Vissink A, Visser A. Dexmedetomidine versus Midazolam in Procedural Sedation. A Systematic Review of Efficacy and Safety. PLoS One. 2017 Jan 20;12(1):e0169525. doi: 10.1371/journal.pone.0169525. eCollection 2017. PMID 28107373
- [Background] Batko I, Koscielniak-Merak B, Tomasik PJ, Kobylarz K, Wordliczek J. Lidocaine as an element of multimodal analgesic therapy in major spine surgical procedures in children: a prospective, randomized, double-blind study. Pharmacol Rep. 2020 Jun;72(3):744-755. doi: 10.1007/s43440-020-00100-7. Epub 2020 Apr 15. PMID 32297162
- [Background] Bellon M, Le Bot A, Michelet D, Hilly J, Maesani M, Brasher C, Dahmani S. Efficacy of Intraoperative Dexmedetomidine Compared with Placebo for Postoperative Pain Management: A Meta-Analysis of Published Studies. Pain Ther. 2016 Jun;5(1):63-80. doi: 10.1007/s40122-016-0045-2. Epub 2016 Feb 10. PMID 26861737
- [Background] Weibel S, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Afshari A, Kranke P. Efficacy and safety of intravenous lidocaine for postoperative analgesia and recovery after surgery: a systematic review with trial sequential analysis. Br J Anaesth. 2016 Jun;116(6):770-83. doi: 10.1093/bja/aew101. PMID 27199310
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743